CLINICAL TRIAL: NCT05661019
Title: Clinical Feasibility of the Myotrace Measurement
Status: Completed | Type: Observational
Sponsor: Philips Clinical & Medical Affairs Global (Industry)
Collaborators: Philips Medizin Systeme (Unknown)
Responsible Party: Sponsor
Other Study IDs: SEF-2023-300047 Myotrace
Record Dates: First submitted 2022-12-13; First posted 2022-12-22 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Respiratory Disease
MeSH Terms: conditions — Respiration Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Obtain Myotrace measurements — Myotrace measurement equipment, consisting of an application (i.e. non-medical software) running on a Philips laptop, Porti7 data acquisition system and software (Twente Medical Systems International (TMSi), Netherlands) (CE-approved), ECG cables, and three standard ECG (for EMG) electrodes. Also an on the shelf accelerometry sensor and respiration belt (TMSi) are used for the NRD measurement (CE-approved).

SUMMARY:
To evaluate the feasibility of the MYOTRACE NRD (Neural Respiratory Drive) index as an aid to assess the respiratory status of a patient (improving or stable versus deteriorating) as compared to a specialist in thoracic medicine's evaluation in a general care setting.

DETAILED DESCRIPTION:
This clinical investigation is designed as a single-arm evaluation of a diseased patient population. This study includes a longitudinal observation study of patients who enter the general ward (admission) until they leave the hospital (discharge).

This study includes standard patient care by the hospital staff with addition of Myotrace measurement, accelerometry and respiratory rate measurement via respiration belt during the NRD measurement.

The primary endpoint of the study is the Neural Respiratory Drive (NRD) index. This index will offline be compared to the specialist in thoracic medicine's assessment of the patient's health status after study closure. The General Ward care team will be blinded to the index values during the study. Re-admission information (i.e. 14 days after discharge) will be collected as well and used in the comparison with NRD index and specialist in thoracic medicine evaluation. Furthermore, the site will be asked to make note of patient events during study participation that are important for the study and study measurements.

The secondary endpoints of the study are the spot-check measurements, other objective and subjective measurements, and the subjective evaluation (e.g. experiences, preferences, acceptance, etc) of the Myotrace measurement protocol/procedures by the healthcare professionals and patients.

In total 50-60 patients will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+, fluent knowledge of English or German.
* Group A: Obstructive ventilatory disorders (conditions resulting in an increased load on the respiratory muscle pump due to hyperinflation ± pronounced hypoxaemia)

  * Acute exacerbation of COPD (pronounced hypoxia OR acute or acute on chronic hypercapnic respiratory failure)
  * Exacerbation of asthma bronchiale
  * Exacerbation of non-CF-bronchiectasis (infectious)
  * Infectious exacerbation of lung disease in cystic fibrosis
* Group B: Conditions with an increase in NRD due to an impairment in gas exchange (particularly die to diffusion limitation and/or ventilation-perfusion-mismatch

  * Exacerbation of an interstitial lung disease (e.g. Idiopathic pulmonary fibrosis (IPF), Non Specific Interstitial Pneumonia (NSIP), Connective tissue disease- associated interstitial lung disease CTD-ILD)
  * Worsening of pulmonary arterial hypertension World Health Organisation (WHO) group 1 (e.g. due decompensated heart failure)
  * Acute pulmonary embolism
  * Pneumonia (resulting in hypoxaemia)

Exclusion Criteria:

* Obesity hypoventilation syndrome (rationale: NRD decreased)
* Obesity WHO III with Body Mass Index (BMI) > 40 kg/m2 (rationale: surface EMG signal quality low)
* Hypercapnic respiratory failure due to hypoventilation of central origin, e.g. opiate-induced, Congenital central hypoventilation syndrome, post stroke (rationale: central respiratory control affected)
* Neuromuscular disease affecting respiratory muscles, e.g. motor neurone disease, muscular dystrophy type Duchenne etc. (rationale: EMG signal quality etc. different)
* Decompensated heart failure with atrial fibrillation (rationale: central breathing disturbance common)
* Patients on chronic opioid therapy (e.g. chronic pain, methadone etc.) (rationale: reduced NRD)
* Self reported pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: During recruitment of the patients, all patients admitted to the general ward who are having a respiratory disease or condition and satisfy the inclusion criteria will be eligible, including patients returning to general ward from ICU admission.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2025-01-09 (Actual); Study Completion 2025-01-09 (Actual)

PRIMARY OUTCOMES:
Evaluate Feasibility of the MYOTRACE NRD index | Mar 2024 (anticipated to be know at end of study)
  to evaluate the feasibility of the MYOTRACE NRD index as an aid to assess the respiratory status of a patient as compared to a specialist in thoracic medicine's evaluation in a general care setting.

SECONDARY OUTCOMES:
Added value of NRD index | Mar 2024 (anticipated to be know at end of study)
  Investigate the added value of the NRD index on patient assessment, in comparison to the other spot-check measures
Assess the viability of the MYOTRACE measurement protocol within the spot check practice | Mar 2024 (anticipated to be know at end of study)
  Assess the viability of the MYOTRACE measurement protocol within the spot check practice
Healthcare/patient satisfaction | Mar 2024 (anticipated)
  Level of healthcare professional as well as patient satisfaction, as captured via semi-quantitative and qualitative survey

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Schwarz, Principal Investigator — University of Zurich
Locations (1):
- University Hospital Zürich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No
All data will stay within Philips. A publication might occur with de-identified patient data.